CLINICAL TRIAL: NCT01255059
Title: GWAS Research of Lung Cancer by Department of Epidemiology and Biostatistics in Tianjin Medical University Cancer Institute and Hospital
Brief Title: GWAS Research of Lung Cancer in Tianjin
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: TMU-CIH-GWASLC-Epi-Tianjin
Record Dates: First submitted 2010-12-05; First posted 2010-12-07 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2012-01

CONDITIONS: Non-small Cell Lung Cancer; Primary Carcinoma
Keywords: Genome-wide association studies(GWAS); Single nucleotide polymorphism(SNP); Lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Peripheral blood sample (10 ml) was collected from each study subject. Buffy coats were isolated and frozen for DNA extraction.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Female lung cancer group: Female, non-smoker, non-small cell lung cancer
- Health control: Female, non-smokers, no lung cancer or other types of cancers' healthy population

SUMMARY:
To study the association of Genetic Polymorphisms with Lung Cancer Risk in Tianjin Population.

DETAILED DESCRIPTION:
Eligibility criteria:

* nonsmoker
* female
* age between 35 and 80
* no other types of tumors history
* frequency-matched cases and controls on gender and age

Outcome measures:

* OR(odds ratio)
* RR(risk ratio)
* CI(confidence interval)
* SAS software

ELIGIBILITY:
Inclusion Criteria:

* Non-small cell lung cancer
* Age from 35 to 80 years old
* Female
* Non-smokers
* Frequency-matched on age and gender

Exclusion Criteria:

* Previous medical history of cancer
* Previous radiotherapy
* Previous chemotherapy

Ages: 35 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients were newly diagnosed and histologically confirmed primary non-small cell lung cancer from Tianjin Medical University Cancer Hospital.The control subjects who underwent health check-up in hospitals were frequency-matched to cases on gender and age. All the subjects were genetically unrelated Chinese with Han ethnicity.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2010-06; Primary Completion 2016-11 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Genetic variant in TP63 on locus 3q28 is associated with risk of lung adenocarcinoma among never-smoking females in Asia | 2011-12
  A GWAS reported a novel association between the TP63 locus and risk of lung adenocarcinoma; however, this association did not achieve genome-wide significance among never-smoking males or females. We genotyped the TP63 SNPs reported by the previous GWAS (rs10937405 and rs4488809) in 500 never-smoking female lung cancer cases and 500 never-smoking female controls from China. Genetic variation in rs10937405 was associated with lung adenocarcinoma. Our findings provide strong evidence that genetic variation in TP63 is associated with risk of lung adenocarcinoma among non-smoking females.

CONTACTS AND LOCATIONS:
Overall Officials: Chen Kexin, M.D., Ph.D, Study Director — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China

REFERENCES:
- [Background] Landi MT, Chatterjee N, Yu K, Goldin LR, Goldstein AM, Rotunno M, Mirabello L, Jacobs K, Wheeler W, Yeager M, Bergen AW, Li Q, Consonni D, Pesatori AC, Wacholder S, Thun M, Diver R, Oken M, Virtamo J, Albanes D, Wang Z, Burdette L, Doheny KF, Pugh EW, Laurie C, Brennan P, Hung R, Gaborieau V, McKay JD, Lathrop M, McLaughlin J, Wang Y, Tsao MS, Spitz MR, Wang Y, Krokan H, Vatten L, Skorpen F, Arnesen E, Benhamou S, Bouchard C, Metspalu A, Metsapalu A, Vooder T, Nelis M, Valk K, Field JK, Chen C, Goodman G, Sulem P, Thorleifsson G, Rafnar T, Eisen T, Sauter W, Rosenberger A, Bickeboller H, Risch A, Chang-Claude J, Wichmann HE, Stefansson K, Houlston R, Amos CI, Fraumeni JF Jr, Savage SA, Bertazzi PA, Tucker MA, Chanock S, Caporaso NE. A genome-wide association study of lung cancer identifies a region of chromosome 5p15 associated with risk for adenocarcinoma. Am J Hum Genet. 2009 Nov;85(5):679-91. doi: 10.1016/j.ajhg.2009.09.012. Epub 2009 Oct 15. PMID 19836008
- [Background] Caporaso N, Gu F, Chatterjee N, Sheng-Chih J, Yu K, Yeager M, Chen C, Jacobs K, Wheeler W, Landi MT, Ziegler RG, Hunter DJ, Chanock S, Hankinson S, Kraft P, Bergen AW. Genome-wide and candidate gene association study of cigarette smoking behaviors. PLoS One. 2009;4(2):e4653. doi: 10.1371/journal.pone.0004653. Epub 2009 Feb 27. PMID 19247474
- [Background] Yoon KA, Park JH, Han J, Park S, Lee GK, Han JY, Zo JI, Kim J, Lee JE, Takahashi A, Kubo M, Nakamura Y, Lee JS. A genome-wide association study reveals susceptibility variants for non-small cell lung cancer in the Korean population. Hum Mol Genet. 2010 Dec 15;19(24):4948-54. doi: 10.1093/hmg/ddq421. Epub 2010 Sep 28. PMID 20876614
- [Background] Rafnar T, Sulem P, Besenbacher S, Gudbjartsson DF, Zanon C, Gudmundsson J, Stacey SN, Kostic JP, Thorgeirsson TE, Thorleifsson G, Bjarnason H, Skuladottir H, Gudbjartsson T, Isaksson HJ, Isla D, Murillo L, Garcia-Prats MD, Panadero A, Aben KK, Vermeulen SH, van der Heijden HF, Feser WJ, Miller YE, Bunn PA, Kong A, Wolf HJ, Franklin WA, Mayordomo JI, Kiemeney LA, Jonsson S, Thorsteinsdottir U, Stefansson K. Genome-wide significant association between a sequence variant at 15q15.2 and lung cancer risk. Cancer Res. 2011 Feb 15;71(4):1356-61. doi: 10.1158/0008-5472.CAN-10-2852. Epub 2011 Feb 8. PMID 21303977